CLINICAL TRIAL: NCT05970731
Title: Directed Topical Drug Delivery for Treatment for PASC Hyposmia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00113299
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-06

CONDITIONS: Post Acute Sequelae Covid-19 Hyposmia
Keywords: Covid-19; smell loss; hyposmia
MeSH Terms: conditions — COVID-19; Anosmia | interventions — Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Beclomethasone (Active Comparator): 84 mcg of Beclomethasone administered twice in each nostril via a microsponge (Day 1 and Day 14)
  Interventions: Drug: Beclomethasone; Device: Microsponge
- Placebo (Placebo Comparator): Placebo (0.9% sodium chloride) administered twice in each nostril via a microsponge (Day 1 and Day 14)
  Interventions: Other: Placebo; Device: Microsponge

INTERVENTIONS:
Drug: Beclomethasone — 84 mcg of Beclomethasone administered topically on an intranasal microsponge, placed in the olfactory cleft using a nasal endoscope, on day 1 and repeated on day 14.
  Arms: Beclomethasone
Other: Placebo — Placebo (0.9% sodium chloride) administered topically on an intranasal microsponge, placed in the olfactory cleft using a nasal endoscope, on day 1 and repeated on day 14.
  Arms: Placebo
Device: Microsponge — Drug delivery using chitosan-based biocompatible microsponge

SUMMARY:
This is a phase II randomized, double-blinded, placebo-controlled study to evaluate the efficacy of topical intranasal treatment of beclomethasone vs. placebo for improved olfactory function.

DETAILED DESCRIPTION:
Eligible participants are randomized to receive either Beclomethasone or placebo intranasally via a microsponge twice on day 1 and day 14. Study duration is three months and includes 4 in-person study visits: 2 visits for drug administration at Baseline and Week 2, and 2 follow-up visits at Week 6 and Week 18. Participants will be expected to complete the Smell Identification Test (SIT) and Questionnaire on Olfactory Disorders (QOD) at baseline, Week 6, and Week 18. The investigator hypothesizes that the application of beclomethasone directly in the nasal cavity will result in improved olfactory function.

ELIGIBILITY:
Inclusion Criteria:

* Post-COVID hyposmia lasting greater than 3 months following COVID19 by history
* Male or female, aged 18 years or older

Exclusion Criteria:

* Pregnancy or lactation
* Known allergic reactions to components of microsponge (including shellfish) or to beclomethasone
* Known diagnosis of glaucoma
* Febrile illness within 1 week
* Treatment with another investigational drug or other intervention within 3 months
* Active sinonasal disease by nasal exam, i.e. rhinosinusitis, nasal polyps
* Adults unable to consent
* Prisoners, employees or subordinates
* Individuals who are not yet adults (infants, children, teenagers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Change in olfactory function as measured by the Smell Identification Test (SIT) | Baseline, 6 weeks, 18 weeks
  The SIT has a score range of 0 to 40, where a higher score reflects better olfactory function.

SECONDARY OUTCOMES:
Change in olfactory quality of life (QOL) measured by the Questionnaire on Olfactory Disorders (QOD) | Baseline, 6 weeks, 18 weeks
  The QOD consists of 17 statements which patients report on a scale of 0 to 3. These scores are summed for a total score range of 0 to 51, where a higher score reflects better olfactory-specific QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Goldstein, MD, PhD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No